CLINICAL TRIAL: NCT07140679
Title: A Phase II Trial of Adjuvant Toripalimab in High Risk Localized Colon Cancer With Mismatch Repair Deficiency
Brief Title: Immunotherapy (Toripalimab) for Reducing Recurrence Risk After Surgery for Mismatch Repair Deficient Stage IIB, IIC, or III Colon Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Coherus Oncology, Inc. (Industry)
Responsible Party: Principal Investigator, Oluwadunni Emiloju, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008833; P30CA138292 (NIH); NCI-2025-05423 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008833 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6483-24 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Localized Colon Carcinoma; Stage IIB Colon Cancer AJCC v8; Stage IIC Colon Cancer AJCC v8; Stage III Colon Cancer AJCC v8
Keywords: immunotherapy; deficient mismatch repair; colon adenocarcinoma; colon cancer; adjuvant therapy; MSI-H colon adenocarcinoma; dMMR colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Biopsy; Specimen Handling; Colonoscopy; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (toripalimab) (Experimental): Eligible consenting participants receive toripalimab intravenously every 3 weeks for 6 months (8 doses) in the absence of disease recurrence or unacceptable toxicity. Following this, patients undergo surveillance follow up with blood tests, computed tomography (CT) scans, colonoscopy at specified intervals until 5 years post-resection. For patients who have a recurrence, a biopsy will be performed at the time of recurrence.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Colonoscopy; Procedure: Computed Tomography; Other: Questionnaire Administration; Drug: Toripalimab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Specimen Collection
Procedure: Colonoscopy — Undergo colonoscopy
Procedure: Computed Tomography — Undergo CT
  Other Names: Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan
Other: Questionnaire Administration — Ancillary studies
Drug: Toripalimab — Given IV
  Other Names: Anti-PD-1 Monoclonal Antibody JS001; JS-001; Loqtorzi; Toripalimab-tpzi

SUMMARY:
This phase II trial tests how well immunotherapy (toripalimab) works for reducing the risk of cancer recurrence after surgery in patients with mismatch repair deficient stage IIB, IIC, or III colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the efficacy of adjuvant toripalimab in patients with resected stage IIB, IIC, and III mismatch repair deficient (dMMR) colon cancer by measuring 3-year disease-free survival.

SECONDARY OBJECTIVES:

I. Define the immune related toxicity profile of toripalimab in the adjuvant setting.

II. Further evaluate the efficacy of adjuvant toripalimab specifically by measuring 3-year relapse free survival (RFS), 5-year disease free survival (DFS), and 5-year overall survival.

TERTIARY/EXPLORATORY OBJECTIVES:

I. To explore immune, ctDNA, and omic markers associated with clinical efficacy (DFS).

II. To assess patient reported outcomes (PRO) and health related quality of life (QoL).

OUTLINE:

Eligible consenting participants will receive toripalimab intravenously every 3 weeks for 6 months (8 doses) in the absence of disease recurrence or unacceptable toxicity. After completion of study treatment, patients are followed up every 6 months until 5 years post-resection. After completion of study medication, participants undergo surveillance follow up with blood tests, computed tomography (CT) scans, colonoscopy at specified intervals until 5 years post-resection. Patient reported outcomes and quality of life will also be assessed with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resected pathologic stage IIB, IIC and III dMMR colon cancer (American Joint Committee on Cancer [AJCC] 8)
* Deficient mismatch repair (MMR) by immunohistochemistry or microsatellite instability (MSI-H) by polymerase chain reaction (PCR) or next generation sequencing (NGS)
* Complete (R0) resection of pathologic stage IIB, IIC and III dMMR colon cancer 4 to 12 weeks prior to first dose of study drug
* Available tissue sample from surgical specimen
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Absolute neutrophil count (ANC) ≥ 1,500 /mcL
* Platelets ≥ 100,000 / mcL
* Hemoglobin ≥ 9 g/dL or ≥ 5.0 mmol/L

  * Transfusion is allowed to obtain an adequate hemoglobin level
* Creatinine ≤ 1.5 x upper limit of normal (ULN) or measured or calculated creatinine clearance ≥ 40 mL/min for patient with creatinine levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance should be calculated per institutional standard
* Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN

  * Patients with previously diagnosed Gilbert syndrome can have total bilirubin < 3.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Signed informed consent
* Patients at least 18 years of age
* Must have had a full colonoscopy prior to enrollment. If synchronous colon cancers are present, both must have deficient MMR and both must have undergone complete resection for patient to be eligible
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment. WOCBP are women younger than 55 years (yrs) of age excluding those who are surgically unable to get pregnant due to prior hysterectomy and or bilateral salpingo-oophorectomy
* Patients of childbearing / reproductive potential should use adequate birth control methods, as defined by the investigator, during the study treatment period and for a period of 90 days after the last dose of study drug. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard
* Female patients who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 90 days after the last dose of study drug

Exclusion Criteria:

* Neoadjuvant treatment for dMMR colon cancer
* Presence of metastatic dMMR colon cancer
* Underlying medical conditions that, in the investigator's opinion, will make the administration of the study drug hazardous or obscure the interpretation of adverse events
* Uncontrolled psychiatric illness or psychological condition potentially hampering compliance with the study protocol and follow-up schedule
* History of pneumonitis requiring treatment with steroids, or history of interstitial lung disease
* History of a hematologic or primary solid tumor malignancy within the last 5 years
* Autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo, diabetes mellitus type 1, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, controlled psoriasis or resolved childhood asthma/atopy not requiring systemic treatment can be enrolled
* Active hepatitis B or hepatitis C
* Systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Treatment with live vaccines within 30 days prior to the first dose of study medication. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, nasal seasonal flu, H1N1 flu, rabies, Bacille Calmette Guerin (BCG) and typhoid vaccine
* Prior treatment with any immune checkpoint inhibitor
* Current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year Disease free survival (DFS) | Time between the date of registration and the first date of documented recurrence or death due to any cause assessed up to 3 years
  Time between the date of registration and the first date of documented recurrence, regardless of discontinuation of study drug, or death due to any cause, assessed at 3 years

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 5 years
  Safety will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. Treatment-related adverse events (defined as potentially, probably and definitely) will be summarized in preferred term by system organ class and listed on an individual subject basis at patient level. Immune-related adverse events will also be tabulated.
3-year Relapse free survival (RFS) | Time between the date of registration and the first date of documented disease recurrence assessed up to 3 years.
  Time between the date of registration and the first date of documented disease recurrence, assessed at 3 years
5-year DFS | Time between the date of registration and the first date of documented recurrence, or death due to any cause assessed up to 5 years
  Time between the date of registration and the first date of documented recurrence, regardless of discontinuation of study drug, or death due to any cause, assessed at 5 years.
Colon cancer specific survival (CCSC) | Time between the date of registration and the date of death due to colon cancer, assessed up to 5 years
  CCSC is the time between the date of registration and the date of death due to colon cancer, assessed up to 5 years
Overall survival (OS) | Time between the date of registration and the date of death due to any cause, assessed up to 5 years
  Time between the date of registration and the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwadunni E. Emiloju, MBBS, MS, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (5):
- United States (5):
  - Emory Decatur Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia